CLINICAL TRIAL: NCT01422460
Title: The Efficacy of Platelets Rich Plasma Injection With PRGF Method in the Treatment for Osteoarthritis of the Subtalar Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC11003011CTIL
Record Dates: First submitted 2011-08-14; First posted 2011-08-24 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Osteoarthritis of Subtalar Joint
Keywords: Osteoarthritis; PRP; PRGF
MeSH Terms: conditions — Osteoarthritis | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet Rich Plasma (Experimental): intra articular injection 2ml of platelet-derived preparation rich in growth factors
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — Platelet Rich Plasma (Preparation Rich in Growth Factors)
  intra articular injection 2ml
  Arms: Platelet Rich Plasma (Preparation Rich in Growth Factors)
  Other Names: Platelet-derived preparation rich in growth factors

SUMMARY:
The investigators will try to find any efficacy of platelet rich plasma injection for the treatment of osteoarthritis (OA) in the subtalar joint. Autologous platelet-secreted growth factors (GFs) may have therapeutic effects in OA capsular joints via multiple mechanisms. The investigators aim is to examine the effect of a platelet-derived preparation rich in growth factors(PRGFs) in OA of the subtalar joint, using parameters of pain, function, quality of life and safety.

DETAILED DESCRIPTION:
The therapeutic use of autologous platelet-rich plasma (PRP) constitutes a relatively new biotechnology that has been a breakthrough in the stimulation and acceleration of soft-tissue and bone healing In this process PRGF (preparation rich in growth factors) combines the advantage of an autologous fibrin clot that will aid in hemostasis as well as provide growth factors in high concentrations to the site of a tissue defect. The platelet-rich plasma preparation encourages the release and slow delivery of growth factors from harvested platelets, activated by endogenous thrombin, and is used as a biological enhancer in the healing of fractures, lumbar fusions, cartilage defects, muscle tears and tendon lesions, thus promoting initiation and early maturation of bone and soft tissue formation which involves a more physiologic repair with less scar tissue.

Few tubes of whole blood are drowning from the patient in a sterile manner and go through a process of centrifugation and laboratory separation of the different plasma fractions. Then, to derive benefit from the described natural mechanism, Ca2+ is added to plasma enriched in platelets, triggering the formation of a fibrin matrix containing embedded platelets. The resulting PRGF allows the slow release of biologically active proteins that initiate and modulate wound healing in both soft and hard tissues .

The objective of this clinical trial is to evaluate the symptomatic efficacy of PRGF application in the treatment of OA of the Sub-Talar joint.

base on that knowledge here is the protocol briefly:

1st visit: Enrollment of patient

1. The patient will be given a full verbal and written explanation regarding the trial and treatment. by the investigator . The patient will sign the informed consent form and will be given a serial number.
2. The screening form :VAS SCORE and ANKLE-HINDFOOT SCORE will be completed-
3. Demographic data: date of birth, sex, age and complete medical history, weight, height and previous treatments will be recorded.
4. Clinical examination will be performed.
5. Blood (4 tubes, 4-5 m"l each) will be drawn from all patients . The blood taken from the PRGF group patients will then be used for the preparation of PRGF.

Intra-Articular injections (PRGF) will then be initiated.

TREATMENT PROCEDURES AND FOLLOW UP VISITS CLINICAL-RADIOLOGICAL ASSESSMENT

* Clinical assessment for all patients shall be made on enrollment, and then 4, 12, 26 weeks after enrollment.
* The clinical assessment will be according to the Ankle- Hindfoot, and the VAS SCORES.
* The radiological evaluation will be according to Kellgren and lawrence and will be performed on AP and Lateral views of the knee.

Side effect will be monitored at every visit

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-70
* Diagnosed OA of subtalar joint
* Patients who didn't benefit from other conservative treatments
* Patients who are willing to participate in the trial

Exclusion criteria:

* Non ambulatory
* Pregnant or lactating women
* Patient with containment disease that may affect joint
* Patient with open wounds; or skin disease; suspected joint infection: in the treated area
* Patients with a specific condition or poor general health status that will interfere with the functional assessments during the study or who had intraarticular injection or have had surgery within the previous 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in function and activity level in subtalar joint with osteoarthritis | 1 year
  function and activity levels -be leveled according to ANKLE HINDFOOT SCORE 1-100
improvement in pain in subtalar osteoarthritis | 1 year
  pain will be leveled according to VAS SCORE:1-10 POINTS (10 THE MOST IN PAIN)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel